CLINICAL TRIAL: NCT03452787
Title: Meta Analysis of Epigenomic and Metabolomic Signatures of APOA2 Gene by Saturated Fat
Brief Title: Epigenomic and Metabolomic Signatures of APOA2 Gene by Saturated Fat Interaction
Status: Completed | Type: Observational
Sponsor: Tufts University (Other)
Responsible Party: Principal Investigator, Jose Ordovas, Senior Scientist, Lab Director JM-USDA-HNRCA, Tufts University
Other Study IDs: APOA2_SATFAT_META_ANALYSIS
Record Dates: First submitted 2018-01-29; First posted 2018-03-02 (Actual); Last update posted 2018-03-02 (Actual); Status verified 2018-03

CONDITIONS: Body Mass Index
Keywords: Body mass index; genetics; diet; saturated fat
MeSH Terms: interventions — Cohort Studies

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Boston Puerto Rican Health Study (NCT01231958): 40 with CC and 40 with TT genotypes at APOA2 rs5082. Participants of each genotype will be further divided into two subgroups based on SFA intake: low, <22 grams/day, high, ≥22 grams/day.
  Interventions: Other: None, cohort studies
- GOLDN (NCT00083369): 107 participants with CC genotype and 272 with TT genotype for APOA2 rs5082.
  Interventions: Other: None, cohort studies
- Framingham Heart Study (NCT00005121): 73 with CC and 170 with TT genotypes at APOA2 rs5082. Participants of each genotype will be further divided into two subgroups based on SFA intake: low, <22 grams/day, high, ≥22 grams/day.
  Interventions: Other: None, cohort studies

INTERVENTIONS:
Other: None, cohort studies — this is a metanalysis of previously obtained observational data. there is not intervention on any of the cohorts.

SUMMARY:
Obesity is driven by genetic and environmental factors. Among the latter, diet is a most important one. The investigators refer to these combinations of genetic and dietary factors as 'gene-diet interactions.' Higher consumption of saturated fats (found mostly in foods of animal origin) has been associated with higher weight in people who were homozygotes for the minor allele at a genetic variant known as APOA2 -265 T>C (rs5082). In the current study, the investigators will seek to gain an understanding of the biological mechanisms driving this interaction. The investigators will select participants in three cohorts according to this genetic factor and conduct a series of molecular analyses (epigenetics, transcriptomics, and metabolomics). The analyses will identify epigenetic marks that are associated with saturated fat intake exclusively in subjects who carry this genetic factor. Moreover, the investigators will examine the association between epigenetic status and genotype at APOA2 and mRNA expression of the gene, and concentrations of metabolites in the blood. This study will increase the understanding of how genetics and diet act together to promote weight gain, and may eventually have implications for dietary recommendations that make use of genetic information.

DETAILED DESCRIPTION:
Background: Apolipoprotein A-II (APOA2) is a significant constituent of high-density lipoproteins (HDL) with an undefined biological role. A putative functional variant, -265 T>C (rs5082) within the APOA2 promoter, has been shown consistently to interact with saturated fat (SFA) intake to influence the risk of obesity.

Objective: This study will implement an integrative approach to characterize the molecular basis of this interaction.

Design: The investigators will conduct an epigenome-wide scan on 80 participants carrying either the rs5082 less common genotype (CC) or the most common genotype (TT) and consuming either a low (<22 g/d) or high (≥22 g/d) SFA diet, matched for age, sex, BMI, and diabetes status in the Boston Puerto Rican Health Study (BPRHS). The investigators then will validate the findings in selected participants in the Genetics of Lipid Lowering Drugs and Diet Network (GOLDN) (n=379) and the Framingham Heart Study (FHS) (n=243). Transcription and metabolomics analyses will be conducted to determine the relationship between epigenetic status, APOA2 mRNA expression, and blood metabolites.

Data sources. The Boston Puerto Rican Health Study (BPRHS), the Genetics of Lipid Lowering Drugs and Diet Network (GOLDN), and the Framingham Heart Study (FHS) Study selection: In BPRHS, 40 participants with CC genotype at APOA2 -265T>C (rs5082) will be selected, with 20 reporting a low SFA intake (<22 g/d) and 20 indicating a high SFA intake (≥22 g/d). By matching age, sex, SFA intake, type 2 diabetes status, and BMI for the 40 participants with CC genotype, the second set of 40 participants with TT genotype of APOA2 -265T>C will be selected from the same population. In GOLDN, 107 participants with CC genotype and 272 with TT genotype for APOA2 -265T>C, who were not taking medication for hypertension, dyslipidemia, or diabetes, will be selected to validate the findings from BPRHS. In FHS, the investigators will include 73 unrelated participants with CC genotype and 170 with TT genotype at APOA2 -265T>C, who did not take medication for hypertension, dyslipidemia, or diabetes. Participants of each genotype will be further divided into two subgroups based on SFA intake: low, <22 grams/day, high, ≥22 grams/day.

Data Extraction. Genome-wide DNA methylation of isolated DNA samples in BPRHS and GOLDN was quantified using Illumina Infinium® human methylation 450K arrays (Illumina, San Diego, CA, USA). The methylation signal at each methylation site will be estimated as a β score, the proportion of total methylation-specific signal, and the detection P-value as the probability that total intensity for a given probe falls within the background signal intensity after normalization and quantity control check. FHS methylome data from dbGaP, accession#:phg000492.v2, where methylation statuses of 2,741 participants were measured in samples taken from participants attending their exam 8 visit between 2005 and 2008, using Illumina Infinium® human methylation 450K array. Methylation signals will be processed and normalized as for BPRHS and GOLDN. The investigators will obtain FHS transcriptome data from dbGaP under accession phe00002.v6. Metabolic profiling of plasma samples from those 80 participants of BPRHS for whom the methylome analysis will be performed by Metabolon, Inc. (Durham, NC, USA) Outcomes: Body mass index will be the only outcome. Data Synthesis. (1) Epigenome-wide analysis of APOA2 genotype, by high and low SFA intake, will be conducted in 80 matched case/control participants of BPRHS, replicated in selected participants of GOLDN, and FHS using linear mixed models. (2) A meta-analysis of the results from the three populations will be conducted using the meta R package.The comparison of allelic effect (beta) of APOA2 -265T>C from the meta-analysis between low and high SFA intake will be conducted with SAS 9.4 using a t-test. (3) Associations between epigenetic variants and APOA2 genotypes with APOA2 mRNA expression will be tested in FHS. (4) Metabolome analysis will be conducted in the same 80 matched case/control participants of BPRHS, and metabolites will be correlated with epigenetic variants at APOA2 locus. (5) Enriched metabolic pathways will be examined in relation to identified epigenetic variants at APOA2 region.

Knowledge translation plan: The results will be disseminated through interactive presentations at local, national, and international scientific meetings and publication in high impact factor journals. Target audiences will include the public health and scientific communities with interest in nutrition, diabetes, obesity, and cardiovascular disease. Feedback will be incorporated and used to improve the public health message and key areas for future research will be defined. Applicant/Co-applicant Decision Makers will network among opinion leaders to increase awareness and participate directly as committee members in the development of future guidelines.

Preliminary findings: In BPRHS, the investigators identified methylation site cg04436964 as exhibiting significant differences between CC and TT participants consuming a high SFA diet, but not among those consuming low SFA. Similar results were observed in GOLDN and FHS. Additionally, in FHS, cg04436964 methylation was negatively correlated with APOA2 expression in participants consuming a high SFA diet. Furthermore, when consuming a high SFA diet, CC carriers had lower APOA2 expression compared to those with the TT genotype, but expression levels were similar when consuming a low SFA diet. Lastly, the metabolomic analysis identified four pathways as overrepresented by metabolite differences between CC and TT genotypes with high SFA intake.

Significance: The investigators will apply multi-omics approaches to investigate the mechanistic foundations of the APOA2 -265T>C genotype by SFA interaction linked to the disruptive condition of obesity. the investigators may uncover plausible dysregulation of several metabolic pathways. This study will illustrate the effectiveness of multiple omics approaches to well-established gene-diet interactions, and contribute new evidence to ongoing explorations of the impact of saturated fat on human health.

ELIGIBILITY:
Inclusion Criteria:

* subjects with the apoA2 genotype TT or CC

Exclusion Criteria:

* all other genotypes

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Individuals extracted from the BPRHS, GOLDN and Framingham Studies
Sampling Method: Probability Sample
Enrollment: 602 (Actual)
Dates: Start 2017-01-01 (Actual); Primary Completion 2017-12-01 (Actual); Study Completion 2017-12-31 (Actual)

PRIMARY OUTCOMES:
Body mass index (BMI) | One time point taken during the first visit of the participants to the studies used for the meta-analyses.
  BMI calculated based on weight (kg) and height (meters) information from each participant using the equation BMI=kg/m2

CONTACTS AND LOCATIONS:
Overall Officials: Jose M Ordovas, PHD, Principal Investigator — JM-USDA-HNRCA at Tufts University
Locations (1):
- JM-USDA-HNRCA at Tufts University, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No
we are getting deidentified data from dbGAP and we cannot shared with any other group

REFERENCES:
- [Background] Delgado-Lista J, Perez-Jimenez F, Tanaka T, Perez-Martinez P, Jimenez-Gomez Y, Marin C, Ruano J, Parnell L, Ordovas JM, Lopez-Miranda J. An apolipoprotein A-II polymorphism (-265T/C, rs5082) regulates postprandial response to a saturated fat overload in healthy men. J Nutr. 2007 Sep;137(9):2024-8. doi: 10.1093/jn/137.9.2024. PMID 17709437
- [Background] Corella D, Peloso G, Arnett DK, Demissie S, Cupples LA, Tucker K, Lai CQ, Parnell LD, Coltell O, Lee YC, Ordovas JM. APOA2, dietary fat, and body mass index: replication of a gene-diet interaction in 3 independent populations. Arch Intern Med. 2009 Nov 9;169(20):1897-906. doi: 10.1001/archinternmed.2009.343. PMID 19901143
- [Background] Smith CE, Ordovas JM, Sanchez-Moreno C, Lee YC, Garaulet M. Apolipoprotein A-II polymorphism: relationships to behavioural and hormonal mediators of obesity. Int J Obes (Lond). 2012 Jan;36(1):130-6. doi: 10.1038/ijo.2011.24. Epub 2011 Mar 8. PMID 21386805
- [Background] Corella D, Tai ES, Sorli JV, Chew SK, Coltell O, Sotos-Prieto M, Garcia-Rios A, Estruch R, Ordovas JM. Association between the APOA2 promoter polymorphism and body weight in Mediterranean and Asian populations: replication of a gene-saturated fat interaction. Int J Obes (Lond). 2011 May;35(5):666-75. doi: 10.1038/ijo.2010.187. Epub 2010 Oct 26. PMID 20975728
- [Background] Corella D, Arnett DK, Tsai MY, Kabagambe EK, Peacock JM, Hixson JE, Straka RJ, Province M, Lai CQ, Parnell LD, Borecki I, Ordovas JM. The -256T>C polymorphism in the apolipoprotein A-II gene promoter is associated with body mass index and food intake in the genetics of lipid lowering drugs and diet network study. Clin Chem. 2007 Jun;53(6):1144-52. doi: 10.1373/clinchem.2006.084863. Epub 2007 Apr 19. PMID 17446329
- [Background] Tucker KL, Mattei J, Noel SE, Collado BM, Mendez J, Nelson J, Griffith J, Ordovas JM, Falcon LM. The Boston Puerto Rican Health Study, a longitudinal cohort study on health disparities in Puerto Rican adults: challenges and opportunities. BMC Public Health. 2010 Mar 1;10:107. doi: 10.1186/1471-2458-10-107. PMID 20193082
- [Background] Lai CQ, Wojczynski MK, Parnell LD, Hidalgo BA, Irvin MR, Aslibekyan S, Province MA, Absher DM, Arnett DK, Ordovas JM. Epigenome-wide association study of triglyceride postprandial responses to a high-fat dietary challenge. J Lipid Res. 2016 Dec;57(12):2200-2207. doi: 10.1194/jlr.M069948. Epub 2016 Oct 24. PMID 27777315
- [Background] DAWBER TR, MEADORS GF, MOORE FE Jr. Epidemiological approaches to heart disease: the Framingham Study. Am J Public Health Nations Health. 1951 Mar;41(3):279-81. doi: 10.2105/ajph.41.3.279. No abstract available. PMID 14819398
- [Derived] Lai CQ, Smith CE, Parnell LD, Lee YC, Corella D, Hopkins P, Hidalgo BA, Aslibekyan S, Province MA, Absher D, Arnett DK, Tucker KL, Ordovas JM. Epigenomics and metabolomics reveal the mechanism of the APOA2-saturated fat intake interaction affecting obesity. Am J Clin Nutr. 2018 Jul 1;108(1):188-200. doi: 10.1093/ajcn/nqy081. PMID 29901700